CLINICAL TRIAL: NCT05453864
Title: Culturally Adapted Manually Assisted Brief Problem-Solving Interventions Plus Trauma-focused Cognitive Behavior Therapy (CMAP Plus TF-CBT) for Suicidal Ideation Among Burn Survivors
Brief Title: CMAP Plus Trauma-focused Cognitive Behavior Therapy for Suicidal Ideation Among Burn Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHAR M- CMAP Plus TFCBT-004
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Suicidal Ideation; Trauma, Psychological
MeSH Terms: conditions — Suicidal Ideation; Psychological Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMAP Plus TFCBT (Experimental): This intervention is a manual-assisted intervention, which will include two existing culturally adapted psychological interventions 1) Culturally Adapted Manual Assisted Psychological (CMAP), 2) Self-help manual for trauma - BASID Ki Kahani. Both interventions are based on the principles of Cognitive behavioural therapy (CBT).
  Interventions: Behavioral: CMAP Plus TFCBT
- Treatment As Usual (TAU) (No Intervention): This will be already receiving local medical, psychiatric and primary care services providing standard routine care to the participants.

INTERVENTIONS:
Behavioral: CMAP Plus TFCBT — This will include 8 individual sessions of CMAP Plus TFCBT delivered by a trained therapist over a period of 12 weeks. Each session will last between 45 to 60 minutes.
  Arms: CMAP Plus TFCBT

SUMMARY:
The study aims to determine whether CMAP Plus TFBCT is feasible and acceptable for burn survivors with suicidal ideations.

To identify any barriers to the recruitment of participants. To determine initial data for the primary outcome measure to perform a sample size calculation for a larger trial.

DETAILED DESCRIPTION:
The study will be conducted in two stages. Stage 1 is to adapt the existing CMAP intervention for burn survivors and integrate it with existing culturally adapted TFCBT intervention. Stage 2 is to test the feasibility and acceptability of study intervention in a Randomised Controlled Trial (RCT).

In the first stage, the adaptation of the intervention will be carried out by a group of experts including bilingual health experts such as psychiatrists and psychologists, the potential users (i.e., burn survivors with Suicidal ideation), and experienced CBT therapists. The expert group will involve in an iterative process of discussion for the adaptation of the intervention including the development of the integrated intervention manual.

Stage 2 will be a rater blind, two-arm, multi-site, feasibility randomized controlled trial (RCT) of CMAP Plus TF CBT for burn survivors with suicidal ideation randomized either to 1) CMAP Plus TF CBT added to Treatment As Usual (TAU) or 2) TAU alone.

A total of N=80 burn survivors with suicidal ideation will be recruited from hospitals (Burn Injuries Units) in Karachi, Lahore, Rawalpindi, Quetta, Peshawar, Multan, and Hyderabad, Pakistan. Each participant in the intervention arm will receive 8 individual sessions of CMAP Plus TFCBT over 12 weeks. Assessment measures will be administered before and after the intervention in the 12th week. All assessments will be rater blind. After post-assessments, a purposefully selected subset (stratified by age & gender) of participants will be invited for qualitative interviews (upto 15) to explore their experiences and satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Had burn injury and identified for having suicidal ideation measures with Beck scale for suicidal Ideation (BSI)
* Able to give informed consent
* Living within the catchment areas of participating hospitals

Exclusion Criteria:

* Unable to provide consent due to severe mental or physical illness
* Unlikely to be available for outcome assessments (temporary residence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility Indicator | From baseline to 12th week (end of intervention)
  The feasibility will be determined by collating data on recruitment and retention rates. The success criterion of feasibility will be to recruit > 50% of eligible participants and retain 70% of participants.
Acceptability Indicator | From baseline to 12th week (end of intervention)
  Intervention acceptability will be assessed using data on attendance. The criterion for acceptability is a mean attendance rate of >70% of sessions. This will also be determined by participant's views on acceptability of intervention content, mode of delivery etc. thorough qualitative interviews.

SECONDARY OUTCOMES:
Beck Scale for Suicide Ideation | From baseline to 12th week (end of intervention)
  This is a 19-item instrument for detecting and measuring the current intensity of the patients' specific attitudes, behaviors, and specificity of a patient's thoughts to kill him/herself during the past week.
The Brief Posttraumatic Growth Inventory | From baseline to 12th week (end of intervention)
  This is a 21-item measure of growth that uses a 6-point Likert-type response scale. It helps to assess individual's growth by using retrospective self-reported items.
Suicide Attempt and Self-Harm | From baseline to 12th week (end of intervention)
  This consists of four questions measuring the previous suicide attempt and the presence of self-harm. The scale was taken from the original Self-Harm Questionnaire
Beck Depression Inventory | From baseline to 12th week (end of intervention)
  This is 21-items scale measuring symptoms of depression. Higher scores on the scale indicate greater severity of depression.
Beck Hopelessness Scale | From baseline to 12th week (end of intervention)
  This instrument is designed to measure three aspects of hopelessness, feelings about the future, loss of motivation and expectations.
The Generalised Anxiety Disorder | From baseline to 12th week (end of intervention)
  This is a 0-3 point rating scale with seven-items to assess common anxiety symptoms of generalised anxiety, panic, social anxiety, and PTSD.
Euro-Qol-5 Dimensions scale | From baseline to 12th week (end of intervention)
  It's a standardised instrument to measure participants' health-related quality of life. It consists of a self-report questionnaire covering five dimensions of health (mobility, self-care, usual activities, pain/ discomfort, and anxiety/ depression)
Problem Solving Inventory | From baseline to 12th week (end of intervention)
  This is one of the most widely used self-report inventories in problem solving.
The coping with burns questionnaire | From baseline to 12th week (end of intervention)
  This scale is to measure coping after discharge from burns unit. Most items in this scale are burn-related and alluded to specific difficulties that burn patients might experience.
Burn Specific Health Scale-Brief | From baseline to 12th week (end of intervention)
  The Burn Specific Health Scale (BSHS) assess burn specific health status of participants.

IPD SHARING:
Plan to Share IPD: No